CLINICAL TRIAL: NCT04512794
Title: Pulmonary Vein Isolation Plus Left Atrial Slow Zone Mapping and Ablation An AcQMap Substrate Characterization Study (PLASZMA)
Brief Title: Pulmonary Vein Isolation Plus Left Atrial Slow Zone Mapping and Ablation
Acronym: PLASZMA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Company decision
Sponsor: Acutus Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CLP-22
Record Dates: First submitted 2020-08-11; First posted 2020-08-14 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Atrial Arrhythmias
Keywords: ablation; atrial arrhythmias

STUDY DESIGN:
Intervention Model Description: The subject population will consist of men and women 18 years of age or older presenting for a de novo ablation of a symptomatic, complex atrial arrhythmia including atrial fibrillation/atrial tachycardia/atrial flutter
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Non-randomized (Other): All subjects with de novo ablation procedure for an atrial arrhythmia using the AcQMap System.
  Interventions: Device: AcQMap High Resolution Imaging and Mapping System

INTERVENTIONS:
Device: AcQMap High Resolution Imaging and Mapping System — Evaluate the safety and effectiveness of the AcQMap System in mapping atrial arrhythmias when a specific procedure work flow is followed.

SUMMARY:
Pulmonary Vein Isolation Plus Left Atrial Slow Zone Mapping and Ablation: An AcQMap Substrate Characterization Study (PLASZMA)

DETAILED DESCRIPTION:
The AcQMap Imaging and Mapping System® is intended for use in patients for whom electrophysiology procedures have been prescribed.

When used with the AcQMap Catheters, the AcQMap System is intended to be used to reconstruct the selected chamber from ultrasound data for purposes of visualizing the chamber anatomy and displaying electrical impulses as either charge density-based or voltage-based maps of complex arrhythmias that may be difficult to identify using conventional mapping systems alone.

AND

When used with specified Patient Electrodes, the AcQMap System is intended to display the position of the AcQMap Catheters and conventional electrophysiology (EP) catheters in the heart.

OR

When used with conventional electrophysiology catheters, the AcQMap System provides information about the electrical activity of the heart and about catheter location during the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age at the time of consent
2. Clinically indicated and scheduled for a de novo catheter ablation of a complex left atrial arrhythmia including AF/AT/AFL
3. Willing and able to provide written informed consent to participate in the study and agree to comply with all follow-up visits and evaluations for the duration of the study.

Exclusion Criteria:

1. In the opinion of the investigator, any contraindication to the planned atrial ablation, including anticoagulation contraindications, renal failure, or sepsis.
2. Atrial arrhythmias secondary to electrolyte imbalance, thyroid disease, or any other reversible or non-cardiac cause.
3. Any DCCV within 60-days of the index procedure where sinus rhythm was not maintained for at least 60-minutes.
4. Any cardiac defibrillator (ICD) or pacemaker implanted within 8-weeks prior to the ablation procedure.
5. History of previous left atrial ablation (including surgical treatment) for AF/AT/AFL.
6. Structural heart disease or cardiac history including:

   1. Left ventricular ejection fraction (LVEF) < 35% based on a 2-d transthoracic echocardiogram (TTE) within the previous 180-days prior to enrollment.
   2. Left atrial size > 60 mm (parasternal long-axis view) based on 2-d TTE within the previous 180-days prior to enrollment.
   3. Prior history of New York Heart Association (NYHA) Class IV heart failure.
   4. Any evidence of NYHA Class III heart failure in the previous 3-months prior to enrollment.
   5. Unstable angina or ongoing myocardial ischemia.
   6. Myocardial infarction (STEMI) within the previous 180-days (sub-endocardial infarct within previous 90-days) prior to enrollment.
   7. Moderate or severe valvular heart disease (stenosis or regurgitation).
   8. Presence of a left atrial appendage occlusion device.
7. Body Mass Index (BMI) > 40kg/m2
8. History of blood clotting or bleeding disease.
9. History of chronic obstructive pulmonary disease (COPD) requiring use of oxygen in the treatment regimen.
10. History of obstructive sleep apnea not currently being treated.
11. Pregnant or lactating (current or anticipated during study follow-up).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Freedom From Device/Procedure Related Major Adverse Events (MAEs) | 6 Months
  MAEs inlcude: death, myocardial infarction, cardiac perforation/tamponade, cerebral infarct, or systemic embolism, Major bleeding requiring transfusion of blood products, Mitral or tricuspid valve damage, Symptomatic pulmonary vein (PV) stenosis, Asymptomatic PV stenosis ≥ 70%, Permanent phrenic nerve injury, Access site complications requiring pharmacological or surgical intervention, Atrio-esophageal fistula, Pericarditis, Heart block requiring a permanent pacemaker, Vagal nerve injury leading to gastroparesis, Other serious adverse device effects (SADEs), including transient ischemic attack (TIAs), adjudicated as "probably or definitely related" to the AcQMap System

SECONDARY OUTCOMES:
Number of Participants Who Experienced at Least One procedure and device related Serious Adverse Events.serious adverse device effects (SADEs), and all unanticipated device effects (UADEs) | 6 Months
  Recording of all SAEs/SADEs/UADEs through 6-months-procedure

OTHER OUTCOMES:
Number of subjects who are free from AF/AT/AFL (following a 90-day blanking period) | 12 Months
  Time to first event of any atrial arrhythmia from day 91 through 12 months.

IPD SHARING:
Plan to Share IPD: No